CLINICAL TRIAL: NCT00230542
Title: Phase II Study of Carboplatin and Pemetrexed in Patients With Recurrent Platinum Sensitive Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Carboplatin and Pemetrexed in Recurrent Platinum Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-220
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: platinum-sensitive recurrence; carboplatin; pemetrexed
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin / Pemetrexed (Experimental): Single Arm Study Carboplatin AUC 5 Pemetrexed 500 mg/m2
  Interventions: Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Carboplatin — Given intravenously following pemetrexed over 30-45 minutes once every three weeks for 6 cycles (18 weeks)
  Other Names: Paraplatin
Drug: Pemetrexed — Given intravenously over 30 minutes once every three weeks for 6 cycles (18 weeks)
  Other Names: Alimta

SUMMARY:
The purpose of this study is to determine the effects (good and bad) the combination of carboplatin and pemetrexed have on patients with recurrent ovarian, peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
* Before patients receive any chemotherapy treatments they will be given three medications to prevent side effects from the chemotherapy drugs. These medications are vitamin B12, folic acid and dexamethasone.
* Chemotherapy treatments will be given intravenously in the outpatient clinic. Pemetrexed will be given first and will take 10 minutes to infuse followed by carboplatin which will take 30-45 minutes to infuse. These treatments will be repeated once every three weeks for 6 cycles of chemotherapy (18 weeks).
* Before each chemotherapy treatment the following tests and procedures will be performed: physical exam and medical history; evaluation of ability to undertake daily activities; and blood tests.
* After every 2 cycles of chemotherapy (every 6 weeks) patients will have a CT or MRI scan to measure how well their cancer is responding to treatment.
* The study treatment will last for 6 cycles of chemotherapy as long as the tumor does not grow and the patient isn't experiencing any severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of platinum-sensitive recurrence of epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* The following histologic subtypes are eligible: papillary serous, endometrioid, mucinous, clear cell, adenocarcinomas, transitional, and mixtures of the above.
* At least one measurable lesion according to RECIST criteria via CT or MRI scan
* Received a platinum-containing regimen at initial diagnosis
* ECOG performance status of 0,1 or 2
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* WBC > 1,500/mm3
* Neutrophils > 1,500/mm3
* Platelets > 100,000/mm3
* Total Bilirubin < 1.5 ULN
* Calculated creatinine clearance > 45 ml/min
* ALT/AST < 3 x ULN (no liver mets) ALT/AST < 5 x ULN (with liver mets)
* Complete recovery from completion of previous chemotherapy or biologic therapy
* Negative pregnancy test and agree to practice effective method of birth control

Exclusion Criteria:

* Patients with sarcomatous, stromal, or germ cell elements
* Prior pelvic radiotherapy > 25% of bone marrow
* Uncontrolled medical problem that in the opinion of the investigator would preclude safe administration of the study drugs
* Past history of bone marrow transplantation or stem cell support
* Known history of CNS metastasis unless the patient has had treatment with surgery or radiation therapy, is neurologically stable, and does not require oral or intravenous corticosteroids or anticonvulsants
* Prior malignancy except adequately treated carcinoma in situ of the uterine cervix, incidental stage I endometrial cancer, basal cell or squamous cell skin cancer or breast cancer (invasive or ductal carcinoma in situ) of which the patient has been disease-free for at least five years
* Routine prophylactic use of G-CSF or GM-CSF or blood transfusions within 2 weeks
* Clinically significant cardiac disease as defined by: history of unstable angina within 6 months; history of symptomatic ventricular arrhythmias; history of congestive heart failure; history of myocardial infarction within 6 months
* Uncontrolled hypercalcemia or diabetes mellitus
* Any signs of intestinal obstruction with bowel function and/or nutrition
* Grade 2 or greater peripheral neuropathy
* Participation in an investigational study within three weeks
* History of anaphylactic shock to prior platinum chemotherapy
* History of psychiatric disability or other central nervous system disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the response rate of carboplatin in combination with pemetrexed in patients with recurrent platinum-sensitive epithelial ovarian cancer, fallopian tube cancer or peritoneal cancer. | 2 years
  This study has now been published: Matulonis U.A.,Horowitz N, Campos S, Lee H., Lee J., Krasner C., Berlin S., Roche M., Duska L, Pereira L, Kendall D, Penson R. Phase II Study of Carboplatin and Pemetrexed for the Treatment of Platinum-Sensitive Recurrent Ovarian Cancer. J Clin Oncol. 2008:26(35):5761-6

SECONDARY OUTCOMES:
To assess time to progression, progression-free survival, and overall survival in this patient population
to assess toxicities of treatment with combination carboplatin and pemetrexed. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts